CLINICAL TRIAL: NCT00748631
Title: Assessment of Percutaneous Balloon Kyphoplasty in the Treatment of Malignant Vertebral Fractures (Multiple Myeloma and Osteolytic Metastases) : "Observational Study"
Brief Title: Treatment of Malignant Vertebral Fractures With Percutaneous Balloon Kyphoplasty.
Acronym: KYPHOK
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the data collected are enough to obtain a qualitative analysis.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P050323
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2014-11

CONDITIONS: Vertebral Fracture; Multiple Myeloma; Osteolytic Metastases
Keywords: Vertebral fracture; Vertebral compression fracture; Multiple Myeloma Bone marrow diseases; Vertebral metastases; Balloon Kyphoplasty
MeSH Terms: conditions — Spinal Fractures; Multiple Myeloma | interventions — Kyphoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): balloon Kyphoplasty
  Interventions: Device: balloon kyphoplasty

INTERVENTIONS:
Device: balloon kyphoplasty — A bilateral approach is chosen to insert working cannulas into the posterior part of the vertebral body through a posterior transpedicular approach.Once inserted, the balloons are inflated using visual, volume and pressure control to create a cavity.The balloons are then deflated and removed. The Bone Filler Device is then advanced through the working cannula towards the anterior part of the cavity and cement is slowly extruded by a stainless steel stylet, acting as a plunger. When the amount of cement from the first Bone Filler Device is delivered in the cavity, it is removed and another Bone Filler Device is advanced through the working cannula.

SUMMARY:
Balloon Kyphoplasty is an alternative to vertebroplasty in the treatment of painful malignant vertebral fractures. This is a mini-invasive percutaneous treatment, aiming to stabilize the vertebral fracture, decrease of pain. This technique also improves patient function. Namely, bedridden patients are often able to resume walking in the days following vertebral cement injection. Advantage of Balloon Kyphoplasty as compared to vertebroplasty is the ability to inject the cement into the diseased vertebral body which shows cortical destruction with lower pressure, thereby possibly reducing cement leakage and related complications.

This is a multicentric, observational prospective study. Patients are evaluated before and after the procedure.

Sixty women or men older than 18 years, with 1 to 3 painful vertebral fracture(s) of malignant origin (due to multiple myeloma or osteolytic vertebral metastasis) will be enrolled. Each patient will be followed during 1 year after the procedure with 7 visits at D-8, D-1, D1, D15, D90, D180, and D360 or until the death of the patient.

The main evaluation outcome is patient self-global satisfaction regarding the procedure on a semi-quantitative satisfaction scale, 15 days after the Balloon Kyphoplasty.

DETAILED DESCRIPTION:
Vertebral compression fractures (VCF) represent an important source of morbidity in patients presenting osteolytic metastatic or myelomatous vertebral involvement. In addition, cancer treatments may induce osteoporosis with an additional risk of vertebral fractures.

* Current medical treatments are symptomatic. They do not treat the fracture itself.
* Vertebroplasty is an interventional radiological technique that consists of injecting, percutaneously, acrylic cement into the fractured vertebra under radiological guidance and local or general anaesthesia, in order to combine two effects: stabilization of the vertebral body fracture and pain reduction.
* Balloon Kyphoplasty is a variant of vertebroplasty which is performed using the KyphX® System (Medtronic., Sunnyvale, California). Balloon kyphoplasty aims at restore vertebral height of the fractured vertebra using an inflatable balloon prior to inject surgical polymethylmetacrylate (PMMA)cement,into the vertebral body to fix the fracture. It is an expensive technique costing around 4,000 euros for up to 2 vertebrae in the same patient. The surgical technique for the procedure has been described by LIBERMEAN et al: A bilateral approach is usually chosen to insert working cannulas into the posterior part of the vertebral body through a posterior transpedicular approach. In case of limited and asymmetric vertebral destruction, a single unilateral approach may be preferred. Fluoroscopy is used to insert the tools and control the procedure. With reaming tools, two working channels are created and the balloons are inserted. The balloons are available in lengths of 10, 15 and 20 mm.

The two balloons (one on each side) should ideally be centered at middle height between the superior and inferior endplates and in the anterior two-thirds of the vertebral body. Balloon placement into the vertebral body is checked using radiopaque markers at the two extremities of the balloon. Once inserted, the balloons are inflated using visual, volume and pressure control to create a cavity. Inflation is stopped when one of the following inflation endpoints is reached: pressure raised over 400 psi, balloon contacts one of the cortical bone of the vertebra or reaching maximal balloon inflation volume. The balloons are then deflated and removed. The mean balloon inflation volume is 2 to 3ml. The Bone Filler Device, filled before with 1.5 ml of PMMA, is then advanced through the working cannula towards the anterior part of the cavity and cement is slowly extruded by a stainless steel stylet, acting as a plunger. When the amount of cement from the first Bone Filler Device is delivered in the cavity, it is removed and another Bone Filler Device is advanced through the working cannula. This step is repeated till a complete fill of the cavity is obtained. The same procedure is repeated through the other working cannula at the contra-lateral pedicle. Filling of the cavity with highly viscous PMMA is performed under continuous fluoroscopic control.

The aim of this study is to quantify the analgesic and patient function improvement of Balloon Kyphoplasty together with complication types and rate in patients with malignant vertebral fractures due to metastatic disease or multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years or older
2. 1 to 3 vertebral compression fracture(s), between T5-L5, responding to the following criteria:

   * at least 15% loss of vertebral body height (anterior, median or posterior);
   * malignant origin (bone metastases, multiple myeloma, hemopathy) assessed by imaging, including an MRI and a CT-SCAN of less than 4 weeks.
   * Pain or painful deterioration less than 3 months old, related to one or more vertebral fractures with a VAS higher than 50/100 mm when changing position, or higher than 40/100 mm if associated with morphine ≥ 30 mg/day ;
3. The pain related to the fractured vertebrae is the more prevalent
4. More than 3 months life expectancy.
5. Blood Platelets rate more than or equal to 50 000/mm3 within the week before balloon kyphoplasty procedure (after a correct blood transfusion).
6. Patient must have signed a consent form.
7. Patient affiliated to social security

Exclusion Criteria:

1. Patient younger than 18
2. Impossibility to perform Balloon Kyphoplasty:

   * Technical impossibility to achieve the percutaneous approach to the vertebra to treat.
   * Vertebral pedicle diameter or height of treated vertebra(e) not sufficient regarding balloon kyphoplasty TROCATHETER size. This should be assessed through prescreening MRI and/or CT-Scan
3. More than three symptomatic vertebral compression fractures in the same vertebral segment.
4. Patient receiving additional local treatment within 15 days after balloon kyphoplasty procedure (surgery, radiofrequency, radiotherapy).
5. Patient with primary bone tumors (eg : osteosarcoma) or single solitary plasmocytoma (patients presenting those tumors on other parts of the body, other than VCF are eligible).
6. Patients presenting sclerotic or mixed vertebral lesions(sclerotic vertebral lesions at another vertebral level are not a contraindication).
7. Patients with less than 3 month life expectancy
8. Patient undergoing an experimental anti-cancerous treatment in Phase I evaluated at the same time
9. Patient having relevant co-morbidities which may interfere with the data management on pain and quality of life.
10. Patient presenting an inadequate vertebra with Balloon Kyphoplasty.
11. Patient undergoing an additional treatment other than balloon kyphoplasty for their vertebral fracture.
12. Patient presenting neurological signs or spinal cord compression or spinal canal narrowing requiring surgical decompression;
13. Patient with a medical or surgical condition not compatible with balloon kyphoplasty procedure (eg : a non-treated local infection)
14. Patient having an allergy to the bone cement and/or to the contrast media used during the balloon kyphoplasty procedure.
15. Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-10; Primary Completion 2009-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients having a residual pain of ≤ 35mm on a VAS scale or a 50 % decrease in daily morphine dose at day 15 after Balloon Kyphoplasty compared to day 0 (day of procedure). | day 15

SECONDARY OUTCOMES:
1° Clinical Outcomes:· Pain evaluation using a visual analogic scale | D-8-D-1, D2 to D5, d15, D90, D180; D360
quality of life evaluation (SF 12). | D-8 to D-1, D2 to D5, D15, D90, D180; D360
Assessment of the pain due to the compression fracture using a VAS scale in the same position as at the inclusion visit (standing or lying down), | D-8 to D-1, D2 to D5, D15, D90, D180; D360
Assessment of the patient global satisfaction score using a LICKERT Scale, | D-8 to D-1, D2 to D5, D15, D90, D180; D360
Percentage of patients who estimate than the pain due to the compression has decreased by more than 50% after the procedure, | day 15
· Percentage of patients who give a positive answer to the following question: "would you agree to undergo a new Balloon Kyphoplasty in case you need it?" | D2 to D5, D15; D90 ; D180; D360
Time elapsed between Balloon Kyphoplasty procedure and patient get up. | D2 to D5; D15;D90
Resumption of the upright position for patients confined to bed due to their vertebral fracture | D2 to D5; D15
Local and general complications related to cement leakage at each vertebral level treated. | each visit
2° Radiological Outcomes: · Modification of the regional kyphosis angle measured by the Traumatic Regional Angle (ART - STAGNARA and NIEDERMANN) for compression fractures of T10 to L5 | D2to dJ5-d15-d90.-d180- d360
Modification of the global Thoracic and lumbar kyphosis angles. | D2 to d5 - D15 - D90 - d180 - d360
3° Therapeutic Outcomes :· Need for radiation at day 30 after Balloon Kyphoplasty in patient presenting with Multiple Myeloma. | D30

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Denis LAREDO, M.D.,PR., Study Director — Assistance Publique - Hôpitaux de Paris; Antoine FEYDY, M.D., PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (4):
- France (4):
  - Hôpital Henri Mondor - Service de Radiologie, Créteil, Val de Marne
  - Hôpital Lariboisière-service de radiologie ostéoarticulaire, Paris
  - Hôpital Cochin - service de radiologie, Paris
  - Hopital Bichat -service de radiologie, Paris